CLINICAL TRIAL: NCT06615531
Title: Effects of Meditation on Human Well Being
Brief Title: Integrating Magnetic Imaging With Rich Phenotypes
Acronym: IMAGINE
Status: Completed | Type: Observational
Sponsor: Tobias Moeller-Bertram (Industry)
Collaborators: Metamorphosis, LLC (Unknown); University of California, San Diego (Other)
Responsible Party: Sponsor-Investigator, Tobias Moeller-Bertram, President, VitaMed Research LLC
Organization: VitaMed Research LLC (Industry)
Other Study IDs: 20211477B
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Intensive Meditation in Novice and Experienced Meditators
Keywords: Meditation; Mind-body interventions; Functional magnetic resonance imaging; Quantitative electroencephalography; Enzyme-linked immunosorbent assay; Metabolome; Proteome; Exosomes; Mystical experiences; Neurite outgrowth; Machine learning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Whole blood
  2. Blood plasma
  3. Buccal cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single group study: Dr Joe Dispenza Week Long Advanced Retreat Attendees
  Interventions: Behavioral: Advanced multi-component meditation practice

INTERVENTIONS:
Behavioral: Advanced multi-component meditation practice — The study intervention is a multi-component advanced guided meditation practice that incorporates elements of focused attention, non-dual, and loving kindness and compassion meditation techniques as well as breathwork components. The practice includes sitting, lying down, standing, and walking components and is carried out at 7-day advanced meditation retreats lead by Joe Dispenza, D.C. These retreats include lecture-based instruction and up to 35 hours of meditation practice.

SUMMARY:
This study will be focused on assessing the molecular, physiological, neuroimaging, and emotional correlates of a week-long intensive meditation retreat experience in a 20-person cohort comprised of healthy participants.

DETAILED DESCRIPTION:
Mind-body interventions including meditation, reconceptualization, and placebo have been shown to improve a broad range of physical and mental health outcomes in both healthy and patient populations. How and what humans think about their health has a significant and quantifiable impact.

Placebo effects, another mind-body technique that creates health improvements, have been shown to impact every major organ system. More recently, open-label placebos, placebos administered without concealment such that the subject is aware of the placebo, have been shown to be effective for a host of health conditions. Open-label placebo effects demonstrate that placebo responses are surprisingly not dependent on deception, positive expectation, or conditioning.

Meditation, yet another mind-body intervention, has been shown to reduce pain, inflammation, stress, anxiety, depression, and to improve immune function, and emotional regulation. Different meditation techniques can produce mystical-type experiences-non-ordinary perceptual, cognitive, and affective states in which the distinction between the perceiver and the perceived is transcended. The specific pathways through which meditation promotes physical and mental health are not yet well understood, but meditation-induced changes in neural activity and on the immune and autonomic nervous systems, as well as meditation-induced molecular changes in gene expression and on the proteome and metabolome suggest that these are both broad and profound.

While each of these mind-body interventions has been studied individually, the combination of meditation, reconceptualization, and open label placebo and their combined effect on health, neural activity, and molecular physiology have never been jointly studied. This exploratory observational study will employ psychometric health questionnaires; functional magnetic resonance imaging (fMRI); quantitative electroencephalography (qEEG); and blood plasma-based real time cell metabolic analysis, quantitative assessment of neurite outgrowth, and high-throughput transcriptomics, proteomics, and metabolomics to investigate the joint neural and biological effects of these three mind-body interventions in a 7-day retreat setting.

ELIGIBILITY:
Inclusion Criteria:

1. Must be 21 years of age or older
2. Must speak English
3. Must be a registered attendee of the advanced week-long meditation retreat
4. Must be in generally good health
5. Must agree to provide blood and buccal samples before and after the retreat
6. Must be willing to wear a Garmin device for the entire retreat
7. Must agree to fMRI scans before and after the retreat
8. Must agree to qEEG measurements before, during, and after the retreat
9. Must complete the research consent in its entirety
10. Must be willing to complete self-report surveys for physical and emotional well-being

Exclusion Criteria:

1. Younger than 21 years of age
2. Non-English speaking
3. Not a registered attendee of the advanced week-long meditation retreat
4. Not willing to complete the research consent
5. Has a serious health condition
6. Not willing to provide blood or buccal samples
7. Does not agree to fMRI scans
8. Not willing to wear a Garmin watch
9. Does not agree to qEEG measurements
10. Not willing or able to complete all self-report surveys

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All study participants are registered for the advanced meditation retreat.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2023-05-06 (Actual); Study Completion 2023-05-06 (Actual)

PRIMARY OUTCOMES:
Functional brain changes as monitored by functional magnetic resonance imaging (fMRI) following an intensive week-long meditation retreat | 1 week
  fMRI scans will be taken on subjects during two conditions (rest and a 15-minute meditation) before and after the week-long retreat to assess changes in brain functional connectivity associated with meditation (meditation vs rest) and resulting from the retreat (pre vs post). It is expected that whole-brain functional connectivity will become more integrated during meditation as well as after the week-long retreat. Resting state network connectivity will be assessed, and it is expected that default mode network (DMN) intra-network connectivity will decrease during meditation and more so post-retreat.
Mystical Experience Questionnaire (MEQ)-30 scores before and after an intensive week-long meditation retreat | 1 week
  Subjects will be given the MEQ-30 survey following a 15-minute scanner meditation before and after the retreat. An increase in MEQ-30 score is indicative of a higher shift in consciousness and presumably to a more favorable psychological state. Scores will be correlated to functional brain changes.
Brain activity changes as assessed by quantitative EEQ (qEEG) before and after an intensive week-long meditation retreat. | 1 week
  Brain scans will be collected by qEEG on all subjects during a 15-minute meditation before and after the retreat to assess brain complexity. It is expected that brain complexity will increase after the week-long retreat.
Blood plasma proteomic and metabolomic analysis before and after an intensive week-long meditation retreat. | 1 week
  An integrative analysis of proteomic and metabolomic expression in blood plasma will be carried out in samples collected before and after the retreat. The expectation is that shifts in biological processes toward an improved state of health will occur after the week-long retreat.

SECONDARY OUTCOMES:
Heart rate variability changes during a week-long meditation retreat | 1 week
  Heart rate data will be collected using a Garmin wristwatch at the beginning of the meditation retreat and continuously throughout the week-long retreat. Beat-to-beat interval data will be used to calculate heart rate variability. Time domain measures will include the mean of R-R intervals (mRR), standard deviation of all R-R intervals (SDRR), root mean square of successive R-R differences (RMSSD), and the percentage of R-R intervals that vary by at least 50 ms (pRR50). Frequency domain measures will include very low frequency (VLF), low frequency (LF), and high frequency (HF) measures.
Effect of meditation-conditioned blood on neurite outgrowth | 1 week
  Human plasma collected before and after the retreat will be used to treat differentiated Phaeochromocytoma 12 (PC12) cells. Live cell imaging will be carried out to quantify neurite outgrowth. The expectation is that meditation-conditioned (post-retreat) plasma will lead to greater neurite outgrowth than unconditioned (pre-retreat) plasma.

OTHER OUTCOMES:
Changes in endogenous opioids after an intensive week-long meditation retreat | 1 week
  The levels of endogenous opioids oxytocin, beta-endorphin, dynorphin, and endogenous cannabinoid anandamide will be measured using enzyme-linked immunosorbent assay (ELISA) in pre- and post-retreat blood plasma samples. The expectation is that one or more of these molecules will be elevated after the week-long meditation retreat.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Moeller-Bertram, MD, Principal Investigator — VitaMed Research LLC
Locations (1):
- VitaMed Research, LLC, Palm Desert, California, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Zeidan F, Martucci KT, Kraft RA, Gordon NS, McHaffie JG, Coghill RC. Brain mechanisms supporting the modulation of pain by mindfulness meditation. J Neurosci. 2011 Apr 6;31(14):5540-8. doi: 10.1523/JNEUROSCI.5791-10.2011. PMID 21471390
- [Background] Ng TKS, Fam J, Feng L, Cheah IK, Tan CT, Nur F, Wee ST, Goh LG, Chow WL, Ho RC, Kua EH, Larbi A, Mahendran R. Mindfulness improves inflammatory biomarker levels in older adults with mild cognitive impairment: a randomized controlled trial. Transl Psychiatry. 2020 Jan 21;10(1):21. doi: 10.1038/s41398-020-0696-y. PMID 32066726
- [Background] Khoury B, Knauper B, Schlosser M, Carriere K, Chiesa A. Effectiveness of traditional meditation retreats: A systematic review and meta-analysis. J Psychosom Res. 2017 Jan;92:16-25. doi: 10.1016/j.jpsychores.2016.11.006. Epub 2016 Nov 18. PMID 27998508
- [Background] Oyler, D. L. et al. The Influence of Meditative Interventions on Immune Functioning: A Meta-Analysis. Mindfulness 14, 1815-1851 (2023).
- [Background] de Castro JM. Meditation has stronger relationships with mindfulness, kundalini, and mystical experiences than yoga or prayer. Conscious Cogn. 2015 Sep;35:115-27. doi: 10.1016/j.concog.2015.04.022. Epub 2015 May 22. PMID 26002763
- [Background] Afonso RF, Kraft I, Aratanha MA, Kozasa EH. Neural correlates of meditation: a review of structural and functional MRI studies. Front Biosci (Schol Ed). 2020 Mar 1;12(1):92-115. doi: 10.2741/S542. PMID 32114450
- [Background] Tang YY, Ma Y, Fan Y, Feng H, Wang J, Feng S, Lu Q, Hu B, Lin Y, Li J, Zhang Y, Wang Y, Zhou L, Fan M. Central and autonomic nervous system interaction is altered by short-term meditation. Proc Natl Acad Sci U S A. 2009 Jun 2;106(22):8865-70. doi: 10.1073/pnas.0904031106. Epub 2009 May 18. PMID 19451642
- [Background] Buric I, Farias M, Jong J, Mee C, Brazil IA. What Is the Molecular Signature of Mind-Body Interventions? A Systematic Review of Gene Expression Changes Induced by Meditation and Related Practices. Front Immunol. 2017 Jun 16;8:670. doi: 10.3389/fimmu.2017.00670. eCollection 2017. PMID 28670311
- [Background] Xue T, Chiao B, Xu T, Li H, Shi K, Cheng Y, Shi Y, Guo X, Tong S, Guo M, Chew SH, Ebstein RP, Cui D. The heart-brain axis: A proteomics study of meditation on the cardiovascular system of Tibetan Monks. EBioMedicine. 2022 Jun;80:104026. doi: 10.1016/j.ebiom.2022.104026. Epub 2022 May 13. PMID 35576643
- [Background] Chen, W. et al. Comprehensive Metabolomic and Lipidomic Analysis Reveals Metabolic Changes After Mindfulness Training. Mindfulness 11, 1390-1400 (2020).